CLINICAL TRIAL: NCT02880332
Title: Endogenous Pain Processing and Effectiveness of Pain Neuroscience Education in Children With Functional Abdominal Pain and Irritable Bowel Syndrome
Brief Title: Pain Processing and Pain Neuroscience Education in Children With Chronic Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Roselien Pas, Dra. Roselien Pas, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AbdominalPainStudy
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Abdominal Pain; Irritable Bowel Syndrome
Keywords: Chronic pain; Endogenous Pain Processing; Central sensitization; Pain neuroscience education
MeSH Terms: conditions — Abdominal Pain; Irritable Bowel Syndrome; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care + Extra care (Active Comparator): This group will receive usual care and one additional session; extra care.
  Interventions: Other: Usual care; Other: Extra care
- Usual care + PNE (Experimental): Next to usual care, this group will also receive pain neuroscience education.
  Interventions: Other: Usual care; Other: Pain Neuroscience education

INTERVENTIONS:
Other: Usual care — During usual care therapy, children and their parents will receive a +/- 1 h session containing bio-medical directed education and information about the gastro-intestinal system and its function. This knowledge will be brought to bear with a hypnotic journey through their body, guided by a nurse with specific expertise in pediatric abdominal pain. Furthermore, the influence of stress on the gastro-intestinal system will be explained, combined with exercises to practise abdominal respiration.
Other: Pain Neuroscience education — This therapy will consist out of a +/- 1 h one-on-one educational session about neurophysiology of pain, adjusted to the child's comprehension status. The content of the education sessions and pictures will be based on the book "Explain Pain" by Butler and Moseley and will include explanation and reassurance about the cause of pain, a brief summary of relevant pain mechanisms and the integral role of psychosocial and physical factors in precipitating and maintaining pain. Metaphors, leaflets, books and audio-visual media will be used in a supportive function to consolidate verbally transmitted information. Parents will participate in the PNE session as well.
  Other Names: PNE
  Arms: Usual care + PNE
Other: Extra care — During this therapy session, all the patient's/ parents questions that arose from the previous session (Usual care) will be answered. Afterwards, the educated content from this previous session will be revised. Nothing new will be taught. At the end of the session, the participant will be asked to demonstrate the previously learned exercises on abdominal respiration. If the exercises are not well performed, the therapist will correct them.
  Arms: Usual care + Extra care

SUMMARY:
The primary scientific objective of the study entails examining whether altered endogenous pain inhibition is present in children with functional abdominal pain (FAP) and irritable bowel syndrome (IBS) compared with healthy controls (Part 1). A secondary objective implies examining whether pediatric pain neuroscience education (PNE) is able to improve pain catastrophizing, pain-related fear, pain intensity (including symptoms and indices of central sensitization) and pain-related functional disability in children with FAP or IBS (Part 2).

DETAILED DESCRIPTION:
Abdominal pain-related functional gastrointestinal disorders (AP-FGIDs) are common in children, showing a prevalence of 13.5% in Western populations and developing countries. Gastrointestinal disorders are categorised within the Rome criteria III, with irritable bowel syndrome (IBS) (65%) and functional abdominal pain (FAP) (35%) as most commonly occurring subtypes, followed by FAP syndrome, functional dyspepsia and abdominal migraine. These numbers call for action, knowing that persistent pain periods associated with AP-FGIDs significantly interferes with a child's daily functioning. Children suffering from AP-FGIDs participate less during recreational activities, show difficulties in maintaining social contacts, are more absent at school and express academic impairments. Additionally, they report decreased health related quality of life and need more health care utilization.

To date, the pathogenesis underlying AP-FGIDs in children remains unclear. Previous studies suggested abnormal brain-gut interaction, altered gut motility, visceral hypersensitivity, psychosocial disturbance and immune activation as possible explanations for the symptoms. In accordance to research in adults with FGIDs evidence is even growing for the contribution of central sensitization (CS) in the development or persistence of AP-FGIDs in children. CS is defined as "an amplification of neural signalling within the central nervous system that elicits pain hypersensitivity" or "increased responsiveness of nociceptive neurons in the central nervous system to their normal or subthreshold afferent input". This process encompasses malfunctioning of descending inhibitory nociceptive pathways which result in dysfunctional endogenous analgesic control and increased activity of descending nociceptive facilitation and overactivity of the pain neuromatrix in the brain. A systematic review addressing the contribution of CS in pediatric chronic pain conditions concluded that manifestations such as somatic hyperalgesia and altered central pain processing in children with recurrent abdominal pain disorders (RAP) and deficient descending inhibitory nociceptive processing in girls with irritable bowel syndrome (IBS) are indicative of CS in some subtypes of AP-FGIDs (review in progress). However, given the heterogeneous study populations, different protocols and methods used to objectify the presence of CS in this review, no clear statement could be made. In addition, no study examining descending inhibitory nociceptive processing in children with FAP was found.

Descending inhibitory nociceptive processing might be dysfunctional in children with FAP and IBS. Anyhow, research demonstrated that this manifestation of CS can be further influenced by the child's characteristics. Behavioural responses, emotional and cognitive aspects are involved in the facilitation of sensitization through an increased cerebral activation of limbic structures, the insula and large areas of the frontal, temporal and parietal cortices, resulting in a diminished inhibition of the descending pathways.

Parental behaviours may also play an important role in the child's adjustment to pain. Parents are considered essential participants in the management of their child's pain, as parental attitudes, responses, and beliefs can influence the child's pain and adherence to treatment. Indeed, both parental solicitous behaviours (e.g., according special privileges to the child) and parental discouraging behaviours (e.g., criticizing the child) have been found to be associated with increased functional disability. Further, evidence suggests that children's own pain beliefs and pain coping skills may be modelled after their parents' (maladaptive) pain beliefs and pain coping skills. Additionally, increased levels of parent emotional distress have been linked to higher levels of child functional disability and self-reported pain. This underscores the importance of including parents in the assessment and treatment of pediatric chronic pain for optimal outcomes.

Negative cognitions of both the parents and the child can develop when they do not understand the origin of the FAP or IBS. Based on the premise that a better understanding of the nature of the illness results in improved patient outcomes, both child and parents should be addressed by education. Given the possible contribution of CS in children with FAP or IBS, education should include explanation and reassurance about the cause of pain, a brief summary of relevant pain mechanisms and the integral role of psychosocial and physical factors in precipitating and maintaining pain. This main content can be given by pain neuroscience education (PNE). PNE has been studied in various adult chronic pain populations and has shown to be effective in changing pain beliefs and improving health status as well as pain coping strategies.

In contrast to a traditional model of tissue injury or nociception and pain, PNE aims to describe how the nervous system interprets information from tissues through peripheral nerve sensitization, central sensitization, synaptic activity and brain processing. It also explains how neural activation, as either upregulation or downregulation, has the ability to modulate the pain experience in response to (or in absence of) nociceptive input. Patients are thus educated that the nervous system's processing of their injury, in conjunction with various psychosocial aspects, determines their pain experience and that pain is not always a true representation of the status of the tissues. Up to recently, no studies have examined the benefits of PNE in the context of pediatric chronic pain. Drawing upon available evidence in adult samples, it is expected that PNE provided to children will lead to beneficial child pain-related outcomes. Involving parents in PNE sessions will facilitate increased parental understanding of biopsychosocial factors that influence their child's pain, as well as learn how they can support their child to manage symptoms.

Concrete, the present study will examine (1) the function of descending inhibitory nociceptive processing in children with FAP or IBS compared to healthy children (Part 1) and whether (2) reconceptualization of pain, by PNE, is able to influence pain catastrophizing, pain-related fear, pain intensity (including symptoms and indices of central sensitization) and pain-related functional disability (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* > 3 months pain
* diagnosis functional abdominal pain or irritable bowel syndrome

Exclusion Criteria:

* Concomitant organic gastrointestinal disease or chronic disease
* Ongoing specific treatment by another health care specialist (physician or psychotherapist) for abdominal pain symptoms
* Previous pain education or relaxation therapy
* Mental retardation
* Insufficient knowledge of the Dutch language
* Preterm birth
* Menstruation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Parent's catastrophic thinking about their child's pain | Change baseline (at recruitment) to post- intervention (1week following intervention), baseline to follow-up (3 weeks following intervention) and post-intervention to follow up (3 weeks following intervention)
  This outcome will be assessed with the Dutch version of the Pain Catastrophizing Scale for Parents (PCS-P) (Goubert et al. 2006). The PCS-P consists of 13 items describing different thoughts and feelings that parents may experience in relation to their child's pain.

SECONDARY OUTCOMES:
Pain intensity (child report) | Baseline (at recruitment), before interventions, 1 week after both interventions and at follow-up (3 weeks following intervention)
  Pain intensity will be measured using the Faces Pain Scale - Revised (FPS-R)(Hicks et al. 2001)(Dutch version), which is a self-report measure of pain intensity developed for children. It contains 6 faces that are presented horizontally. Children will be asked to point to the face that best reflects the intensity of their current pain and their pain over the last week (average, highest and lowest).
Pain-related fear (parent report) | Baseline (at recruitment), before interventions, 1 week after both interventions and at follow-up (3 weeks following intervention)
  For parental report, the Parent Fear of Pain Questionnaire (PFOPQ)(Simons et al. 2015) will be used. The PFOPQ assesses a parent's fears and avoidance behaviours associated with their child's pain. For child report, the Kuttner Anxiety Scale will be used. This measure consists of faces for assessing pain-related fear even in young children. A Dutch translation will be used for both measures.
Functional disability (parent proxy report) | Baseline (at recruitment), before interventions, 1 week after both interventions and at follow-up (3 weeks following intervention)
  The Functional Disability Inventory (FDI)(Dutch version)(Crombez et al. 2003) is a parent-report inventory for children that measures perceived difficulty in physical and psychosocial functioning due to physical health. It consists of 15 items to be rated on a five-point scale (0-4) concerning perceptions of activity limitations during the past 2 weeks. Total scores range from 0 to 60. Higher scores indicate greater disability.
Pain-related fear (child report) | Baseline (at recruitment), before interventions, 1 week after both interventions and at follow-up (3 weeks following intervention)
  For child report, the Kuttner Anxiety Scale will be used. This measure consists of faces for assessing pain-related fear even in young children. A Dutch translation will be used for both measures.
Hyperalgesia | Baseline (at recruitment) and at follow-up (3 weeks following last intervention)
  Hyperalgesia will be assessed by evaluating pressure pain thresholds (PPT) at a symptomatic test site (rectus abdominus near the umbilical region) and two remote test sites (tibialis anterior and trapezius) with a hand-held pressure Algometer (Wagner Instruments, FPX 25).
Endogenous pain inhibition | Baseline (at recruitment) and at follow-up (3 weeks following last intervention)
  Within the CPM paradigm the perceived pain intensity to a test stimulus before and during/after the addition of a harmful conditioning stimulus will be measured. This study will use the Cold Pressure Task as 'conditioning stimulus' and mechanical stimulation to perform a 'test stimulus'.

CONTACTS AND LOCATIONS:
Overall Officials: Roselien Pas, MSc, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfven G. The pressure pain threshold (PPT) of certain muscles in children suffering from recurrent abdominal pain of non-organic origin. An algometric study. Acta Paediatr. 1993 May;82(5):481-3. doi: 10.1111/j.1651-2227.1993.tb12727.x. PMID 8518526
- [Background] Brown LK, Beattie RM, Tighe MP. Practical management of functional abdominal pain in children. Arch Dis Child. 2016 Jul;101(7):677-83. doi: 10.1136/archdischild-2014-306426. Epub 2015 Dec 23. PMID 26699533
- [Background] Caes L, Vervoort T, Eccleston C, Goubert L. Parents who catastrophize about their child's pain prioritize attempts to control pain. Pain. 2012 Aug;153(8):1695-1701. doi: 10.1016/j.pain.2012.04.028. Epub 2012 May 31. PMID 22657401
- [Background] Crombez G, Bijttebier P, Eccleston C, Mascagni T, Mertens G, Goubert L, Verstraeten K. The child version of the pain catastrophizing scale (PCS-C): a preliminary validation. Pain. 2003 Aug;104(3):639-646. doi: 10.1016/S0304-3959(03)00121-0. PMID 12927636
- [Background] Duarte MA, Goulart EM, Penna FJ. Pressure pain threshold in children with recurrent abdominal pain. J Pediatr Gastroenterol Nutr. 2000 Sep;31(3):280-5. doi: 10.1097/00005176-200009000-00015. PMID 10997373
- [Background] Goubert L, Eccleston C, Vervoort T, Jordan A, Crombez G. Parental catastrophizing about their child's pain. The parent version of the Pain Catastrophizing Scale (PCS-P): a preliminary validation. Pain. 2006 Aug;123(3):254-263. doi: 10.1016/j.pain.2006.02.035. Epub 2006 Apr 27. PMID 16644128
- [Background] Hermann C, Zohsel K, Hohmeister J, Flor H. Cortical correlates of an attentional bias to painful and innocuous somatic stimuli in children with recurrent abdominal pain. Pain. 2008 Jun;136(3):397-406. doi: 10.1016/j.pain.2008.01.007. Epub 2008 Feb 13. PMID 18276076
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Jackson T, Pope L, Nagasaka T, Fritch A, Iezzi T, Chen H. The impact of threatening information about pain on coping and pain tolerance. Br J Health Psychol. 2005 Sep;10(Pt 3):441-51. doi: 10.1348/135910705X27587. PMID 16238858
- [Background] Korterink JJ, Diederen K, Benninga MA, Tabbers MM. Epidemiology of pediatric functional abdominal pain disorders: a meta-analysis. PLoS One. 2015 May 20;10(5):e0126982. doi: 10.1371/journal.pone.0126982. eCollection 2015. PMID 25992621
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] McMurtry MC. How do I love thee? Let me count the ways of responding and regulating. Pain. 2014 Aug;155(8):1421-1422. doi: 10.1016/j.pain.2014.05.011. Epub 2014 May 15. No abstract available. PMID 24837845
- [Background] Meeus M, Nijs J. Central sensitization: a biopsychosocial explanation for chronic widespread pain in patients with fibromyalgia and chronic fatigue syndrome. Clin Rheumatol. 2007 Apr;26(4):465-73. doi: 10.1007/s10067-006-0433-9. Epub 2006 Nov 18. PMID 17115100
- [Background] Merskey, H. & Bogduk, N., 1994. IASP Task Force on Taxonomy Part III: Pain Terms, A Current List with Definitions and Notes on Usage. IASP Task Force on Taxonomy, pp.209-214. Available at: http://www.iasp-pain.org/Content/NavigationMenu/GeneralResourceLinks/PainDefinitions/default.htm#Pain.
- [Background] Millan MJ. Descending control of pain. Prog Neurobiol. 2002 Apr;66(6):355-474. doi: 10.1016/s0301-0082(02)00009-6. PMID 12034378
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Moseley GL. Evidence for a direct relationship between cognitive and physical change during an education intervention in people with chronic low back pain. Eur J Pain. 2004 Feb;8(1):39-45. doi: 10.1016/S1090-3801(03)00063-6. PMID 14690673
- [Background] Moshiree B, Zhou Q, Price DD, Verne GN. Central sensitisation in visceral pain disorders. Gut. 2006 Jul;55(7):905-8. doi: 10.1136/gut.2005.078287. PMID 16766744
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162
- [Background] Van Oosterwijck J, Meeus M, Paul L, De Schryver M, Pascal A, Lambrecht L, Nijs J. Pain physiology education improves health status and endogenous pain inhibition in fibromyalgia: a double-blind randomized controlled trial. Clin J Pain. 2013 Oct;29(10):873-82. doi: 10.1097/AJP.0b013e31827c7a7d. PMID 23370076
- [Background] Palermo TM, Chambers CT. Parent and family factors in pediatric chronic pain and disability: an integrative approach. Pain. 2005 Dec 15;119(1-3):1-4. doi: 10.1016/j.pain.2005.10.027. Epub 2005 Nov 18. No abstract available. PMID 16298492
- [Background] Roth-Isigkeit A, Thyen U, Stoven H, Schwarzenberger J, Schmucker P. Pain among children and adolescents: restrictions in daily living and triggering factors. Pediatrics. 2005 Feb;115(2):e152-62. doi: 10.1542/peds.2004-0682. PMID 15687423
- [Background] Schoth DE, Georgallis T, Liossi C. Attentional bias modification in people with chronic pain: a proof of concept study. Cogn Behav Ther. 2013;42(3):233-43. doi: 10.1080/16506073.2013.777105. Epub 2013 Jun 4. PMID 23731349
- [Background] Seifert F, Maihofner C. Central mechanisms of experimental and chronic neuropathic pain: findings from functional imaging studies. Cell Mol Life Sci. 2009 Feb;66(3):375-90. doi: 10.1007/s00018-008-8428-0. PMID 18791842
- [Background] Sieberg CB, Williams S, Simons LE. Do parent protective responses mediate the relation between parent distress and child functional disability among children with chronic pain? J Pediatr Psychol. 2011 Oct;36(9):1043-51. doi: 10.1093/jpepsy/jsr043. Epub 2011 Jul 8. PMID 21742755
- [Background] Staud R, Craggs JG, Robinson ME, Perlstein WM, Price DD. Brain activity related to temporal summation of C-fiber evoked pain. Pain. 2007 May;129(1-2):130-42. doi: 10.1016/j.pain.2006.10.010. Epub 2006 Dec 6. PMID 17156923
- [Background] Turk DC, Okifuji A. Psychological factors in chronic pain: evolution and revolution. J Consult Clin Psychol. 2002 Jun;70(3):678-90. doi: 10.1037//0022-006x.70.3.678. PMID 12090376
- [Background] Vervoort T, Trost Z, Sutterlin S, Caes L, Moors A. Emotion regulatory function of parent attention to child pain and associated implications for parental pain control behaviour. Pain. 2014 Aug;155(8):1453-1463. doi: 10.1016/j.pain.2014.04.015. Epub 2014 Apr 21. PMID 24769189
- [Background] Vervoort T, Huguet A, Verhoeven K, Goubert L. Mothers' and fathers' responses to their child's pain moderate the relationship between the child's pain catastrophizing and disability. Pain. 2011 Apr;152(4):786-793. doi: 10.1016/j.pain.2010.12.010. Epub 2011 Jan 26. PMID 21272996
- [Background] Vervoort T, Logan DE, Goubert L, De Clercq B, Hublet A. Severity of pediatric pain in relation to school-related functioning and teacher support: an epidemiological study among school-aged children and adolescents. Pain. 2014 Jun;155(6):1118-1127. doi: 10.1016/j.pain.2014.02.021. Epub 2014 Mar 12. PMID 24631587
- [Background] Vervoort T, Caes L, Trost Z, Sullivan M, Vangronsveld K, Goubert L. Social modulation of facial pain display in high-catastrophizing children: an observational study in schoolchildren and their parents. Pain. 2011 Jul;152(7):1591-1599. doi: 10.1016/j.pain.2011.02.048. Epub 2011 Apr 2. PMID 21459512
- [Background] Wilder-Smith CH, Schindler D, Lovblad K, Redmond SM, Nirkko A. Brain functional magnetic resonance imaging of rectal pain and activation of endogenous inhibitory mechanisms in irritable bowel syndrome patient subgroups and healthy controls. Gut. 2004 Nov;53(11):1595-601. doi: 10.1136/gut.2003.028514. PMID 15479679
- [Background] Williams AE, Heitkemper M, Self MM, Czyzewski DI, Shulman RJ. Endogenous inhibition of somatic pain is impaired in girls with irritable bowel syndrome compared with healthy girls. J Pain. 2013 Sep;14(9):921-30. doi: 10.1016/j.jpain.2013.03.003. Epub 2013 May 17. PMID 23685184
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Youssef NN, Atienza K, Langseder AL, Strauss RS. Chronic abdominal pain and depressive symptoms: analysis of the national longitudinal study of adolescent health. Clin Gastroenterol Hepatol. 2008 Mar;6(3):329-32. doi: 10.1016/j.cgh.2007.12.019. Epub 2008 Feb 7. PMID 18258491
- [Background] Heymen S, Maixner W, Whitehead WE, Klatzkin RR, Mechlin B, Light KC. Central processing of noxious somatic stimuli in patients with irritable bowel syndrome compared with healthy controls. Clin J Pain. 2010 Feb;26(2):104-9. doi: 10.1097/AJP.0b013e3181bff800. PMID 20090435
- [Derived] Pas R, Meeus M, Malfliet A, Baert I, Oosterwijck SV, Leysen L, Nijs J, Ickmans K. Development and feasibility testing of a Pain Neuroscience Education program for children with chronic pain: treatment protocol. Braz J Phys Ther. 2018 May-Jun;22(3):248-253. doi: 10.1016/j.bjpt.2018.02.004. Epub 2018 Mar 4. PMID 29550259